CLINICAL TRIAL: NCT02263326
Title: Dolutegravir Antiretroviral Strategy to Promote Improvement and Reduce Drug Exposure (ASPIRE) Study
Brief Title: Dolutegravir Antiretroviral Strategy to Promote Improvement and Reduce Drug Exposure
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Babafemi Taiwo (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Babafemi Taiwo, Professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASPIRE
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dolutegravir plus lamivudine (Experimental): dolutegravir 50 mg plus lamivudine 300 mg once daily
  Interventions: Drug: dolutegravir; Drug: lamivudine
- Continue current ART regimen (Active Comparator): Continue current DHHS recommended or alternative three-drug antiretroviral regimen
  Interventions: Drug: Continue current antiretroviral regimen

INTERVENTIONS:
Drug: dolutegravir — 50 mg tablet by mouth once daily for 48 weeks
  Other Names: TIVICAY, DTG
  Arms: dolutegravir plus lamivudine
Drug: lamivudine — 300 mg tablet by mouth once daily for 48 weeks
  Other Names: EPIVIR, 3TC
  Arms: dolutegravir plus lamivudine
Drug: Continue current antiretroviral regimen — Continue current DHHS recommended or alternative three-drug antiretroviral regimen
  Arms: Continue current ART regimen

SUMMARY:
HIV-1 infected subjects with CD4 nadir > 200 cells/mm3, no history of virologic failure and plasma HIV RNA <50 copies/mL for at least 48 weeks while on any United States Department of Health and Human Services (DHHS) recommended or alternative three-drug antiretroviral regimen will be randomized to dolutegravir (DTG) plus lamivudine (Arm 1) or continuation of their current regimen (Arm 2) for 48 weeks. The primary endpoint is virologic failure defined as confirmed plasma HIV-1 RNA > 50 copies/mL before or at Week 24

DETAILED DESCRIPTION:
DESIGN HIV-1 infected subjects with CD4 nadir > 200 cells/mm3, no history of virologic failure and plasma HIV RNA <50 copies/mL for at least 48 weeks while on any United States Department of Health and Human Services (DHHS) recommended or alternative three-drug antiretroviral regimen will be randomized to dolutegravir (DTG) plus lamivudine (Arm 1) or continuation of their current regimen (Arm 2) for 48 weeks. The primary endpoint is virologic failure defined as confirmed plasma HIV-1 RNA > 50 copies/mL before or at Week 24

All subjects will undergo routine monitoring including plasma HIV-1 RNA, CD4/CD8 count, hematology, chemistry and fasting lipids. Resistance testing will be done in all patients who experience virologic failure. Single-copy HIV-1 assay will be done to quantify residual viremia.

DURATION 48 weeks

SAMPLE SIZE 90 subjects

POPULATION HIV-1-infected men and women, 18 years and older, with CD4 nadir > 200 cells/mm3, no baseline resistance, no history of virologic failure, and HIV RNA <50 copies/mL for at least 48 weeks prior to study entry while on any DHHS recommended or alternative three-drug regimen

REGIMEN Subjects will be randomized (1:1) to:

Arm 1: dolutegravir 50 mg plus lamivudine 300 mg once daily OR Arm 2: Continue current DHHS recommended or alternative three-drug antiretroviral regimen

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infection
* HIV-1 RNA <50 copies/mL on all measurements within 48 weeks prior to study entry while on any DHHS recommended or alternative three-drug antiretroviral regimen. (A history of switching for simplification and/or tolerability is allowed. At least two measurements within the previous 48 weeks are required prior to study screening.)
* No history of virologic failure, defined as consecutive HIV RNA > 50 copies/mL after 12 months of initiating ART. An isolated (non-consecutive) HIV RNA > 50 copies/mL (but less than 400 copies/mL) is permitted after 12 months of initiating ART but not in the 48-week window prior to study entry.
* Screening plasma HIV RNA < 20 copies/mL using the COBAS AmpliPrep/COBAS TaqMan HIV-1 Test V2.0, obtained within 45 days prior to study entry
* Nadir CD4 count >200 cells/mm
* Pretreatment genotype documenting no mutations in the protease or reverse transcriptase genes
* No known resistance to integrase inhibitors
* Laboratory values obtained within 45 days prior to study entry:

ANC >750 Hemoglobin >10 g/dL Platelets >50,000 Calculated creatinine clearance (CrCl) >50 mL/min

* Negative serum or urine pregnancy test
* Men and women age greater or equal to 18 years.
* Ability to continue current regimen (i.e, have uninterrupted access)
* No evidence of chronic hepatitis B

Exclusion Criteria:

* Serious illness or AIDS-related complication within 21 days of screening requiring systemic treatment and/or hospitalization
* Treatment within 30 days prior to study entry with immune modulators
* Vaccination within 7 days
* Active HCV treatment or anticipated need for treatment within study period. (HCV infection alone is not exclusionary)
* Unstable liver disease or severe hepatic impairment
* Known allergy or hypersensitivity to DTG or lamivudine.
* Active drug or alcohol use or dependence that could interfere with adherence to study requirements
* ALT (alanine aminotransferase) >5 x ULN (upper limit of normal) OR ALT >3 x ULN and total bilirubin >1.5 x ULN (with 35% direct bilirubin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babafemi Taiwo, MBBS, Principal Investigator — Northwestern University
Locations (7):
- United States (7):
  - University of California San Diego, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cornell University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Taiwo BO, Marconi VC, Berzins B, Moser CB, Nyaku AN, Fichtenbaum CJ, Benson CA, Wilkin T, Koletar SL, Colasanti J, Acosta EP, Li JZ, Sax PE. Dolutegravir Plus Lamivudine Maintains Human Immunodeficiency Virus-1 Suppression Through Week 48 in a Pilot Randomized Trial. Clin Infect Dis. 2018 May 17;66(11):1794-1797. doi: 10.1093/cid/cix1131. PMID 29293895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Started | 44 | 45
Completed | 43 | 44
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [37 to 56] | 50 [41 to 53] | 47 [38 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 39 | 39 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 35 | 40 | 75
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 15 | 34
  White | 23 | 29 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
CD4 Cell Count [Median (Inter-Quartile Range); unit: cells/mm3] | 694 [533 to 1034] | 646 [380 to 819] | 680 [498 to 927]
Time on Antiretroviral Therapy [Median (Inter-Quartile Range); unit: years] | 5.28 [3.81 to 7.49] | 6.03 [3.72 to 7.44] | 5.7 [3.72 to 7.48]
Current ART Regimen [Count of Participants; unit: Participants]
  Integrase Inhibitor | 18 | 15 | 33
  Protease Inhibitor | 14 | 15 | 29
  Nonnucleoside reverse transcriptase inhibitor | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment Failure
Description: Proportion of participants with treatment failure (defined as virologic failure (HIV RNA >50 copies/mL), loss to follow-up, or treatment discontinuation) between those who switch to DTG + lamivudine and those who continue their current ART regimen
Time Frame: 24 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 44 | 45
proportion of participants | 0.0682 | 0.0667
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; A sample size of 41 participants per arm provided 80% power to show noninferiority of DTG/3TC to cART based on a 12% noninferiority margin, assuming an estimated treatment failure rate of 5% per arm by week 24 and 5% 1-sided type I error rate; Test type: Non-Inferiority — We considered DTG/3TC was noninferior to cART if the 90% confidence interval for the difference in proportions, calculated with Miettinen-Nurminen (score) confidence limits, excluded the 12% noninferiority margin; Risk Difference (RD) = 0.0015, 90% CI 2-sided [-0.098 to 0.102]

2. Secondary Outcome: Proportion of Participants With Virologic Success
Description: Proportion of participants with virologic success (<50 copies/mL) based on FDA snapshot definition
Time Frame: 48 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 44 | 45
proportion of participants | 0.9091 | 0.8889
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Non-Inferiority — The difference in virologic outcomes based on the FDA snapshot algorithm at week 48 (HIV RNA <50 copies/mL) was compared between arms, with 95% confidence intervals; Risk Difference (RD) = 0.020, 95% CI 2-sided [-0.126 to 0.165]

3. Secondary Outcome: Change in CD4 Count From Baseline to Week 48
Description: Change in CD4 count between arms will be presented in the attached statistical analysis table
Time Frame: Baseline and 48 weeks
Population: Population with CD4 count data available at baseline and week 48
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 40 | 43
cells/mm^3 | 39 [-71 to 188] | 28 [-36 to 83]
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Other; p = 0.866, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 48
Description: Change in Total Cholesterol between arms will be presented in the attached statistical analysis table
Time Frame: Baseline and 48 weeks
Population: Population with total cholesterol data available at baseline and week 48
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 40 | 43
mg/dL | 0 [-31 to 31] | -1 [-13 to 9]
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Other; p = 0.613, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in LDL Cholesterol From Baseline to Week 48
Description: Change in Low-density lipoprotein (LDL) cholesterol between arms will be presented in the attached statistical analysis table
Time Frame: Baseline and Week 48
Population: Population with LDL cholesterol data available at baseline and week 48
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 40 | 43
mg/dL | 2 [-19 to 27] | -3 [-16 to 10]
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Other; p = 0.420, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Creatinine Clearance From Baseline to Week 48
Description: Change in Creatinine Clearance between arms will be presented in the attached statistical analysis table
Time Frame: Baseline and Week 48
Population: Population with creatinine clearance data available at baseline and week 48
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 41 | 43
ml/min | -4 [-14 to 4] | 0 [-6 to 5]
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Other; p = 0.074, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Drug Resistance Associated Mutations
Description: Drug resistance mutations measured by HIV genotyping in patients with confirmed virologic failure
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 44 | 45
Participants | 0 | 0

8. Other Pre Specified Outcome: Residual Viremia by HIV-1 Single-copy Assay
Description: Difference in HIV-1 detection by the HIV-1 single copy assay between arms will be presented in statistical analysis
Time Frame: 48 weeks
Population: Participants with HIV-1 single copy assays performed at baseline and week 48 timepoints
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
Number analyzed (Participants) | 36 | 36
copies/mL | 4.7 (7.0) | 4.2 (6.0)
Statistical Analysis 1: Comparison: Dolutegravir Plus Lamivudine vs Continue Current ART Regimen; Test type: Other; p = 0.76, Regression, Linear; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-3.0 to 4.1]

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: After study entry, all laboratory values greater than or equal to Grade 3, any laboratory values that lead to a change in study treatment, and all renal, liver function tests, and lipid values, regardless of grade, were reported. All Grade ≥3 signs/symptoms, any signs/symptoms regardless of grade that lead to a change in treatment, or that meet Expedited Adverse Event (EAE), SAE, or ICH guidelines.
Arm/Group | Dolutegravir Plus Lamivudine | Continue Current ART Regimen
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/44 | 2/45
Other Adverse Events (participants affected / at risk) | 0/44 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolutegravir Plus Lamivudine (N=44) | Continue Current ART Regimen (N=45)
Grade 4 viral syndrome (Infections and infestations) | 1 (1) | 0 (0)
Grade 4 myocardial infarctions (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolutegravir Plus Lamivudine (N=44) | Continue Current ART Regimen (N=45)
Grade 3 bilirubinemia (Hepatobiliary disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02263326/Prot_SAP_ICF_000.pdf